CLINICAL TRIAL: NCT04221529
Title: Single-Arm Phase II-Study in Patients With Extensive Stage Small Cell Lung Cancer (ES-SCLC) With Poor Performance Status Receiving Atezolizumab-Carboplatin-Etoposide
Brief Title: Patients With ES-SCLC and ECOG PS=2 Receiving Atezolizumab-Carboplatin-Etoposide
Acronym: SPACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-TRK-0119
Record Dates: First submitted 2019-09-12; First posted 2020-01-09 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: SCLC, Extensive Stage
Keywords: Atezolizumab
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab (Experimental): Four 21-day cycles of induction therapy with atezolizumab+carboplatin+etoposide followed by 21-day cycles of maintenance therapy with atezolizumab.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg i.v. on day 1 of each cycle

SUMMARY:
Small cell lung cancer (SCLC) is a rapidly proliferating, neuroendocrine tumor that accounts for about 15% of all lung cancers. Most patients have metastases at primary diagnosis involving sites like bone, adrenal glands, liver and brain.

Compared with non-small-cell lung cancer (NSCLC) SCLC has a unique natural history with a shorter doubling time, higher growth fraction, earlier development of widespread metastases, and uniform initial response to chemo- or radiotherapy.

The combination of cis- or carboplatin and etoposide is the standard of care in the first-line treatment of stage IV (extensive-disease) SCLC (ED-SCLC). Despite response rates of 50-80%, most patients relapse within six months and the median survival time is less than 10 months. Between 14 and 23% of SCLC patients develop brain metastases.

New cytotoxic agents as well as targeted therapies have not been able to show any improvement of survival in this group of patients.

Early phase trials of PD 1/PD L1-blocking immunotherapeutic agents in patients with recurrent or ED SCLC have shown promising response rates and good tolerability. Immunotherapy may also contribute to the efficacy of systemic treatment by maintaining initial responses to chemotherapy. A double-blind, placebo-controlled phase 3 trial indicates that the addition of atezolizumab to standard chemotherapy significantly improves overall survival and progression-free survival compared with chemotherapy alone in treatment-naïve patients with ED-SCLC who are in good general condition (ECOG 0 or 1). However, about one in three SCLC patients has a poor performance status (ECOG≥2), which is associated with even shorter survival times of under eight months. At present, there is little information regarding the feasibility, safety and efficacy of adding atezolizumab to standard chemotherapy for this considerable fraction of patients.

The investigators expect, that atezolizumab in addition to chemotherapy is feasible in patients with stage IV SCLC and reduced performance status and therefore crucial efficacy data can be acquired in this trial to evaluate a putative Phase III transition in this particular patient population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent including participation in translational research obtained from the subject prior to performing any protocol-related procedures, including screening evaluations that are not SOC.
* ECOG 2
* At least one measurable tumor lesion (according to RECIST1.1)
* Histologically confirmed small cell lung cancer (SCLC)
* Stage IV disease (according to UICC8)
* No active autoimmune disease
* Adequate organ function defined as:

  * neutrophil count > 1.5 x 109/L
  * thrombocytes ≥ 100 x 109/L
  * hemoglobin ≥ 9 g/dL
  * INR ≤ 1.4 or aPTT ≤ 40 sec during the last 7 days before therapy [Subjects under therapeutic anticoagulation are permitted.]
  * bilirubin < 1.5 x ULN
  * AST (SGOT)/ALT (SGPT) < 3 x institutional ULN (< 5 x ULN in case of liver metastases)
  * creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 45 mL/min
* Availability of tumor tissue/block
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the first dose of IMP.
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. [WOCBP should use an adequate method to avoid pregnancy for 6 months after the last dose of IMP.]
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving IMP and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 6 months after the last dose of IMP. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile) and men who are azoospermic do not require contraception.
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow-up.

Exclusion Criteria:

* Any preceding systemic anticancer therapy for stage IV SCLC. [Up to one full-cycle-dosing of carboplatin+etoposide chemotherapy within the context of SOC is permitted prior to study treatment.] (Note: Prior treatment for limited stage disease allowed).
* Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lives of previously used trial medication, whichever is longer
* Prior therapy with an anti-Programmed cell death protein 1 (anti-PD-1), anti-Programmed cell death-ligand 1 (anti-PD-L1), anti-Programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor [TNFR] family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Previous treatment in the present study (does not include screening failure).
* Symptomatic CNS metastases. [Patients with asymptomatic brain metastases may be included.]
* Major surgery ≤ 28 days before first dose of study treatment
* Any uncontrolled systemic disease, condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results, including but not limited to:

  1. known active HBV, HCV or HIV infection [Patients who are HIV-positive are allowed in the trial, so long as they are stable on anti-retroviral therapy, have a CD4 count ≥ 200 cells/μL, and have an undetectable viral load at the time of screening.]
  2. active tuberculosis
  3. any other active infection requiring systemic therapy
  4. history of allogeneic tissue/solid organ transplant
  5. diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of IMP
  6. other active malignancy requiring treatment
  7. clinically significant or symptomatic cardiovascular/cerebrovascular disease (incl. myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) within 6 months before enrolment
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year).
* Known hypersensitivity to carboplatin, etoposide or atezolizumab or any of the constituents of the product.
* Medication that is known to interfere with any of the agents applied in the trial.
* Any condition or disease which might interfere with the subject's ability to comply with the study procedures (e.g., dementia).
* Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities [§ 40 Abs. 1 S. 3 Nr. 4 AMG].
* Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | Measured from first dose of experimental IMP (or first dose of chemotherapy, whichever occurs first) through study completion, an average of one year.
  OS is defined as the length of time from first dose of experimental IMP (or first dose of chemotherapy, whichever occurs first) to the date of death. A subject who has not died will be censored at last known date alive.

SECONDARY OUTCOMES:
Objective response rate (ORR) (RECIST 1.1) | Starting from Screening up to an average of one year.
  ORR is defined as the proportion of All Treated Subjects whose best overall response (BOR) from baseline is either a CR or PR per RECIST 1.1 criteria. BOR is determined by the best response designation recorded between the base-line assessment (must precede the date of first dose of IMP) and the date of objectively documented progression. For subjects without documented progression, all available response designations will contribute to the BOR determination. Among All Treated Subjects the ORR (based on investigator assessments according to RECIST 1.1) will be summarized by binomial response rates and their corresponding two-sided 95% exact CIs using Clopper-Pearson method.
Progression-free suvival (PFS) | Starting from Screening up to an average of one year.
  PFS is defined as the time from first dose of IMP to the date of the first documented tumor progression, based on investigator assessments (per RECIST 1.1), or death due to any cause.
Incidence of Treatment-Emergent adverse events, serious adverse events and laboratory abnormalities leading to treatment discontinuation | Starting from Screening up to an average of one year.
  The incidence of treatment-emergent adverse events, serious adverse events and laboratory abnormalities leading to treatment discontinuation will be used as an indicator for safety and tolerability of the IMP. Toxicities in these incidents will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Quality of life (EORTC-QLQ-C30) | Starting from Screening up to an average of one year.
  QoL questionnaires (EORTC-QLQ-C30, i.e. European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaire with 30 questions for patients with cancer) will be analyzed according to the respective recommendations and manuals (scoring and interpretation materials) issued by the creators of the instruments.
  Patients have to answer 28 questions from "not at all" (1) to "very much" (4), where lower scores mean a better outcome. The last two questions range from "very poor" (1) to "excellent" (7), where higher scores mean a better outcome.
Quality of life (PRO-CTCAE) | Starting from Screening up to an average of one year.
  QoL questionnaires (PRO-CTCAE, i.e. Patient Reported Outcome - Common Terminology Criteria for Adverse Events) will be analyzed according to the respective recommendations and manuals (scoring and interpretation materials) issued by the creators of the instruments.
  Patients have to answer 22 questions either ranging from "none", "mild", "moderate", "severe" to "very severe" or from "not at all", "a little bit", "somewhat", "quite a bit" to "very much". Lower values mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Reck, Prof. Dr., Principal Investigator — LungenClinic Grosshansdorf
Locations (19):
- Austria (3):
  - Klinikum Klagenfurt, Klagenfurt
  - Universitätsklinikum Krems, Krems
  - Karl Landsteiner Institut für Lungenforschung und Pneumologische Onkologie c/o Wilhelminenspital der Stadt Wien, Vienna
- Germany (16):
  - St. Josef Hospital, Bochum
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Niels-Stensen-Kliniken, Georgsmarienhütte
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - Asklepios Klinik Altona, Hamburg
  - Universität Heidelberg, Heidelberg
  - Klinikum Löwenstein gGmbH, Löwenstein
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Johannes Wesling Klinikum, Minden
  - Klinikum der Universität München, München
  - Brüderkrankenhaus St. Josef, Paderborn
  - Fachkliniken Wangen, Wangen
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
  - Helios Universitätsklinikum, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de
- See also: AIO-Studien-gGmbH — http://www.aio-studien-ggmbh.de